CLINICAL TRIAL: NCT01334905
Title: A Phase 1, Open-Label, Single Oral Dose Study to Assess the Safety, Pharmacokinetics and Effect of Food on the Pharmacokinetics of Mirabegron (YM178) in Healthy Volunteers
Brief Title: A Study to Investigate the Safety and Effect of Food on the Pharmacokinetics of YM178 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Taiwan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 178-CL-092
Record Dates: First submitted 2011-04-12; First posted 2011-04-13 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2011-10

CONDITIONS: Healthy Volunteer; Pharmacokinetics of YM178
Keywords: Overactive Bladder; Urinary incontinence; YM178; mirabegron; Food effect
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A group (Experimental): fasted condition then fed condition
  Interventions: Drug: YM178
- Part B group (Experimental): fed condition then fasted condition
  Interventions: Drug: YM178

INTERVENTIONS:
Drug: YM178 — oral
  Other Names: mirabegron

SUMMARY:
The purpose of the study is to evaluate safety of YM178 and the effect of food intake on the pharmacokinetics of YM178 in healthy adult subjects.

DETAILED DESCRIPTION:
A open-label, randomized, crossover study to assess the effect of food on the pharmacokinetics of single dose of YM178 administered under fasted and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* A normal or clinically non-significant 12 lead ECG as well as normal or clinically non-significant laboratory test results at the time of Screening
* Body weigh at least 50 kg in male and 45 kg in female and body mass index (BMI) between 18.5 and 26.9 kg/m2
* All women of child bearing potential are required to use adequate contraception consisting of two forms of birth control

Exclusion Criteria:

* Hypersensitivity to YM178 or other beta-3 agonists or any of the constituents of the formulation used
* Liver function test values above the upper limit of normal
* A history or presence of psychiatric illness, serious active or recurrent infection
* A previous history of cancer other than basal cell carcinoma or Stage 1 squamous cell carcinoma that has not been in remission for at least 5 years prior to the study
* Donated or lost ≥ 500 mL blood within 3 months or donated plasma within 2 weeks prior to the study
* Receiving or being anticipated to receive a prescription drug or OTC medications within 14 days prior to the study
* Consuming alcohol, xanthine derivative-containing food/beverages (tea, chocolate), grapefruit juice, grapefruit-containing products or Seville oranges (e.g., bitter marmalade) within 48 hours before the study
* A history of substance abuse, drug addiction, or alcoholism within past 2 years prior to the study
* currently participating in another clinical trial or taking or has been taking an investigational drug at least 60 days

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of YM178 | Up to 96 hrs post dose
AUC (area under the curve) of YM178 plasma concentration | Up to 96 hrs post dose

SECONDARY OUTCOMES:
tmax of YM178 plasma concentration | Up to 96 hrs post dose
t1/2 of YM178 plasma concentration | Up to 96 hrs post dose
Safety assessed by the incidence of adverse events, clinical lab tests, vital signs, 12-lead ECGs and physical exam. | Up to 96 hrs post dose

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Taipei, Taiwan